CLINICAL TRIAL: NCT06860789
Title: A Phase I Study to Assess the Safety, Tolerability, Pharmacokinetics, and Preliminary Efficacy of AK135 for the Treatment of Chemotherapy-Induced Peripheral Neuropathy (CIPN) in Patients With Malignant Tumors
Brief Title: AK135 in Patients With Chemotherapy-Induced Peripheral Neuropathy (CIPN)
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Akeso (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: AK135-101
Record Dates: First submitted 2025-02-25; First posted 2025-03-06 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-02

CONDITIONS: Chemotherapy-induced Peripheral Neuropathy (CIPN)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AK135 (Experimental): Each subject will receive a single dose of AK135 every 2-week cycle (Q2W) or every 1-week cycle (QW) or every 3-week cycle (Q3W).
  Interventions: Drug: AK135

INTERVENTIONS:
Drug: AK135 — IV infusion, specified dose with specified treatment frequency

SUMMARY:
A Phase I open label, dose-escalation and expansion study to evaluate the safety, tolerability, pharmacokinetics and preliminary efficacy of AK135 for the treatment of chemotherapy-induced peripheral neuropathy in patients with malignant tumor

ELIGIBILITY:
Inclusion Criteria:

1. Written and signed informed consent.
2. Eastern Cooperative Oncology Group (ECOG) Performance Score of 0 or 1.
3. Life expectancy ≥ 3 months.
4. Histologically or cytologically documented malignant tumor.
5. Previous anti-tumor therapy causing peripheral neurotoxicity that has been discontinued for at least 1 month before enrollment.
6. Diagnosed with Chemotherapy-Induced Peripheral Neuropathy (CIPN) by an oncologist or neurologist, with at least grade 2 NCI Common Terminology Criteria for Adverse Events.
7. Must have pain and/or numbness due to chemotherapy-induced peripheral neuropathy (CIPN) symptoms.
8. Adequate organ function.

Exclusion Criteria:

1. Pharmacologic or non-pharmacologic treatment for CIPN within 2 weeks before the first dose of AK135.
2. Concurrent and/or scheduled to start any anti-tumor treatment that may cause Chemotherapy-Induced Peripheral Neuropathy (CIPN) within 3 months after the first dose of AK135.
3. Concurrent and/or scheduled to start any anti-tumor treatment that may cause hand-foot skin reaction within 3 months after the first dose of AK135.
4. Presence with other illnesses may result in peripheral neuropathy including, autoimmune diseases, diabetes and metabolic syndrome, peripheral vascular disease, infections, nerve injury or compression, vitamin deficiencies, and so on.
5. Skin lesions may affect the assessment of peripheral neuropathy.
6. Unresolved toxicities from prior anti-cancer therapy within 2 weeks before the first dose of AK135, defined as not having resolved to NCI CTCAE v5.0 Grade 0 or 1, or levels specified in the inclusion/exclusion criteria, except for alopecia, and neuropathy.
7. Known allergy or reaction to any component of the AK135 formulation. History of severe hypersensitivity reactions to other mAbs.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Estimated)
Dates: Start 2025-02-28 (Estimated); Primary Completion 2026-03-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Adverse events | From time ICF is signed until 90 days after last dose of AK135
  Incidence and severity of participants with adverse events
DLT | During the first treatment cycle of AK135 （14 days）

SECONDARY OUTCOMES:
EORTC-QLQ-CIPN20 | through study completion, an average of 12 weeks
  Patient-assessed European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-CIPN twenty-item scale
BPI-SF | through study completion, an average of 12 weeks
  Patient-assessed Brief Pain Inventory-Short Form
CTCAE-Neuropathy | through study completion, an average of 12 weeks
  Physician-assessed Common Terminology Criteria for Adverse Events-Neurotoxicity
Cmax of AK135 | through study completion, an average of 12 weeks
AUC | through study completion, an average of 12 weeks
t1/2 | through study completion, an average of 12 weeks
ADAs | From first dose of study drug through 30 days after last dose of study drug.
  Number of subjects who develop detectable anti-drug antibodies

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Sun Yat-sen Memorial Hospital, Guangzhou
  - Shanghai GoBroad Cancer Hospital, Shanghai